CLINICAL TRIAL: NCT07140835
Title: A Prospective Crossover Study Evaluating the Pedal-Controlled Surgistep Platform to Improve Ergonomics in Neurosurgical Operations
Brief Title: Evaluation of the Pedal-Controlled Surgistep Platform to Improve Ergonomics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Atman Desai, Clinical Professor, Stanford University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 80476
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SurgiStep Platform (Experimental): The surgeon will be performing the surgery by standing over the SurgiStep Platform. The duration of the usage depends on the length of the surgery being performed by the surgeon. Surgeons will be using this platform for 2 weeks, after which they will be operating on standard foot stool for 2 weeks.
  Interventions: Device: SurgiStep Platform; Device: Standard Foot stool
- Standard surgical practice (Placebo Comparator): The surgeon will be performing the surgery by standing over the standard of care (foot stool). The duration of the usage depends on the length of the surgery being performed by the surgeon. Surgeons use standard foot stool for 2 weeks, and switch to SurgiStep platform for 2 weeks.
  Interventions: Device: SurgiStep Platform; Device: Standard Foot stool

INTERVENTIONS:
Device: SurgiStep Platform — The Surgistep (pedal-controlled, adjustable platform) allows real-time height adjustment during surgery. The surgeons can adjust the height of the platform.
Device: Standard Foot stool — Foot stool is considered as the standard of care during surgery.

SUMMARY:
Primary Aim: Assess improvement in ergonomics and musculoskeletal discomfort with the Surgistep compared to a standard footstool.

ELIGIBILITY:
Inclusion Criteria:

* Regularly perform neurosurgical procedures (cranial/spine)
* Willing to use both devices (multiple times each).

Exclusion Criteria:

* Severe MSK conditions preventing device usage
* Inability/refusal to participate in observation or surveys.

Ages: 36 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rapid Entire Body Assessment (REBA) Scale Score | During the surgery upto 60 minutes
  The REBA (Rapid Entire Body Assessment) score, used to assess the risk of musculoskeletal disorders (MSDs) in work tasks, ranges from 1 to 15. A lower REBA score indicates a lower risk, with scores below 4 considered to have minimal risk. Higher scores indicate increased risk, with scores of 8 or more indicating a high risk that requires immediate attention and intervention
Rapid Upper Limb Assessment (RULA) Scale Score | During the surgery upto 60 minutes
  The RULA (Rapid Upper Limb Assessment) scale ranges from 1 to 7, with lower scores indicating lower risk and higher scores indicating higher risk of musculoskeletal disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Atman Desai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No